CLINICAL TRIAL: NCT05670678
Title: Improved Respiratory Infection Outcomes Associated With Lactoferrin Fortified a2 Growing up Formula Consumption in Children of 2 to 3 Year Old: a Randomized, Open Label Trial
Brief Title: Improved Respiratory Infection by Consuming Lactoferrin Fortified a2 Growing up Formula in Children of 2 to 3 Year Old
Status: Completed | Type: Observational
Sponsor: a2 Milk Company Ltd. (Industry)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 22-SM-11-A2-001
Record Dates: First submitted 2022-12-20; First posted 2023-01-04 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Infection; Diarrheal Disease
Keywords: growing up stage 3 formula; lactoferrin; acute respiratory infection; diarrheal disease
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- a2 growing up stage 3 formula puls lactoferrin supplement: per 100g serving
  * Lactoferrin 30 mg
  * Galactooligosaccharides (GOS) at 3 g
  * DHA 0.37
  * Lactoferrin supplement plus: 2.68 ml per serving, 20 mg per 2 ml, 600 mg per bottle
  Interventions: Dietary Supplement: a2 growing up stage 3 formula puls lactoferrin supplement
- Enfinitas growing up stage 3 formula: per 100g serving
  * Lactoferrin 330 mg
  * Galactooligosaccharides (GOS) at 1.58 mg
  * β-Glucan 22 mg
  * DHA 0.4
  Interventions: Dietary Supplement: Enfinitas growing up stage 3 formula

INTERVENTIONS:
Dietary Supplement: a2 growing up stage 3 formula puls lactoferrin supplement — The participants in this group will consume 4-5 scoops (8.5g/scoop) of the assigned formula each time, and 4 times per day
  Groups: a2 growing up stage 3 formula puls lactoferrin supplement
Dietary Supplement: Enfinitas growing up stage 3 formula — The participants in this group will consume 4 scoops (10g/scoop) of the assigned formula each time, and 3 times per day
  Groups: Enfinitas growing up stage 3 formula

SUMMARY:
The goal of this observational study is to compare the incidence of ARI and/or diarrheal disease associated with feeding different formulas with and without lactoferrin supplement in children of 2-3 years old. 200 children eligible for the study will be enrolled from two study sites and randomly assigned to two groups (a2 growing up stage 3 formula puls lactoferrin supplement, and Enfinitas growing up stage 3 formula) to feed for 90 days. About 160 children (80 for each group) are expected to finish the study, and data will be collected during the four visits across the study.

Researchers will compare the two groups to see if there is significant decrease of the occurrence of diarrheal disease and/or acute respiratory infection for children fed with a2 growing up stage 3 formula puls lactoferrin supplement

DETAILED DESCRIPTION:
This study is two arms, opening parallel-designed, observational study. Diarrheal and infectious episodes, including acute upper and lower respiratory infections (ARI), changes in stool patterns, use of systemic antibiotics, adverse events and study formula consumption will be compared in children 2 - 3 years of age who are assigned to receive one of the two following study formulas for a 3-month feeding period: a2 growing up stage 3 formula puls lactoferrin supplement and Enfinitas growingup stage 3 formula.

200 children eligible for the study will be enrolled from two study sites and randomly assigned to two groups to feed for 90 days. About 160 children (80 for each group) are expected to finish the study, and data of primary and secondary outcomes will be collected during the four visits across the study. A sample size of 80 completed per group is needed to achieve a 80% power.

The Andersen-Gill model will be used to model the primary outcome (recurrent event of either diarrheal disease or an acute respiratory infection) under the framework of the proportional hazard assumption. For other secondary outcomes such as duration of acute respiratory infections(ARI) and/or diarrheal disease, episodes of systemic antibiotic use,amount of study formula consumed,changes in stool pattern and cost of treatment will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Full term born children current aged 2-3 years old
* Birth weight not less than 2500g (5lb 8oz)
* Consumes Milk or milk-based beverage regularly before recruitment
* Informed consent signed
* Parents or guardians of the infants committ not to participate in interventional clinical research during the intervention

Exclusion Criteria:

* Has a potential risk of metabolic or chronic disease; Fetal malformation; Or present with condition(s) that the investigator believes may affect the infant's ability to be orally fed, the infant's normal growth/development, or the infant's health evaluation.
* In-take prebiotics or probiotic continuesly 15 days before the recruitment.
* Growth problems or other protencial risks.
* Larger-gestational age (LGA) babies born to mothers with gestational diabetes (defined as newborns whose birth weight is above the 90th percentile of average - Treated with antibiotics 7 days before study intervention.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full term born children who are 2-3 years old and consume Milk or milk-based beverage regularly
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Change of frequency of acute respiratory infection (ARI) and/or diarrheal disease | baseline day 0, day 90
  Change of frequency of acute respiratory infection (ARI) and/or diarrheal disease from baseline to 3 months

SECONDARY OUTCOMES:
Duration of acute respiratory infections(ARI) and/or diarrheal disease | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Number of days with acute respiratory infections(ARI) and/or diarrheal disease for each visit
Number of days of antibiotics treated | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Number of days of antibiotics treated for each visit interval
Amount of study formula consumed | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Amount of study formula consumed (in grams)
Changes in stool pattern | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Average number of bowel movements per week and stool consistency
Cost of medical treatment | baseline day 0, visit 1 day 30, visit 2 day 60, visit 4 day 90
  Cost of medical treatment in RMB yuan for each visit interval

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Sheng, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Nan Quan Community Hospital, Jinhua, Zhejiang
  - Qiu Bin Community Hospital, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li F, Jin X, Liu B, Zhuang W, Scalabrin D. Follow-up formula consumption in 3- to 4-year-olds and respiratory infections: an RCT. Pediatrics. 2014 Jun;133(6):e1533-40. doi: 10.1542/peds.2013-3598. Epub 2014 May 19. PMID 24843061
- [Background] Leyer GJ, Li S, Mubasher ME, Reifer C, Ouwehand AC. Probiotic effects on cold and influenza-like symptom incidence and duration in children. Pediatrics. 2009 Aug;124(2):e172-9. doi: 10.1542/peds.2008-2666. Epub 2009 Jul 27. PMID 19651563
- [Background] Gibson GR, Roberfroid MB. Dietary modulation of the human colonic microbiota: introducing the concept of prebiotics. J Nutr. 1995 Jun;125(6):1401-12. doi: 10.1093/jn/125.6.1401. PMID 7782892
- [Background] Boehm G, Lidestri M, Casetta P, Jelinek J, Negretti F, Stahl B, Marini A. Supplementation of a bovine milk formula with an oligosaccharide mixture increases counts of faecal bifidobacteria in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2002 May;86(3):F178-81. doi: 10.1136/fn.86.3.f178. PMID 11978748
- [Background] Cheng JB, Wang JQ, Bu DP, Liu GL, Zhang CG, Wei HY, Zhou LY, Wang JZ. Factors affecting the lactoferrin concentration in bovine milk. J Dairy Sci. 2008 Mar;91(3):970-6. doi: 10.3168/jds.2007-0689. PMID 18292252